

**Sponsor**: CicloMed **Protocol**: CPX-POM-001

Statistical Analysis Plan (TFL shells):

| | SPONSOR: CicloMed |
|----------|-----------------------------------------|
| | PROTOCOL NUMBER: |
| | CPX-POM-001 |
| ST | ATISTICAL ANALYSIS PLAN<br>(TFL shells) |
| Author: | |
| Version: | Version 1.0 |
| Date: | 02FEB2018 |



**Sponsor**: CicloMed **Protocol**: CPX-POM-001

Statistical Analysis Plan (TFL shells):

Version 1.0 / 02FEB2018

### **Cover and signature pages**

| Sponsor: | CicloMed |
|---|---|
| Protocol Number: | CPX-POM-001 |
| Study Title: | A Phase 1, First-in-Human, Safety, Dose Tolerance, Pharmacokinetics, and Pharmacodynamics Study of CPX-POM in Patients with Advanced Solid Tumors |
| Document Version No | Version 1.0 |

We, the undersigned, confirm that we have read, understood and agree to the content of this document and hereby authorise its approval.

| Name Title, Organisation | Signature | Date |
|--------------------------|-----------|------|



(TFL shells):


### **Table of Contents**

| COVER AND SIGNATURE PAGES | 2 |
|---|---|
| Table 14.1-1 – Patients disposition (All patients) | |
| Table 14.1-2 – Number (%) of Patients in the Analysis Populations (All patients) | 12 |
| Table 14.1-3 – Summary of Demography (ITT Population) | 13 |
| Table 14.1-4 – Protocol Deviations (Safety Population) | 18 |
| Table 14.1-5.1 – Disease Characteristics (Safety Population) | 19 |
| Table 14.1-5.2 – Other Medical History (Safety Population) | 21 |
| Table 14.1-6.1.1 – Prior Medications by Therapeutic Class and Preferred Term (Safety Population) | 23 |
| Table 14.1-6.1.2 – Concomitant Medications by Therapeutic Class and Preferred Term (Safety Population) | 24 |
| Table 14.1-7 – Overall Exposure to Study Drug and Drug Compliance (Safety Population) | 25 |
| Table 14.2.1 – Patients who have had at least one other post-baseline tumor assessment (Efficacy Population) | 26 |
| Table 14.2.2 – Summary of Patients Responses (Efficacy Population) | 27 |
| Table 14.3-1.1 – Overview of Adverse Events (Safety Population) | 29 |



(TFL shells):

| Table 14.3-1.2 – Number (%) of Patients with Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) |
|---|
| Table 14.3-1.3 – Number (%) of Patients with Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population)3 |
| Table 14.3-1.4 – Number (%) of Patients with Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) |
| Table 14.3-1.5 – Number (%) of Patients with Serious Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population)3 |
| Table 14.3-1.6 – Number (%) of Patients with Treatment-Emergent Adverse Events Leading to Discontinuation by System Organ Class and Preferred Term (Safety Population) |
| Table 14.3-1.7 – Number (%) of Patients with Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Maximal Severity (Safety Population)3 |
| Table 14.3-1.8 – Number (%) of Patients with Related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Maximum Severity (Safety Population) |
| Table 14.3-1.9 – Number (%) of Patients with Treatment-Emergent Adverse Events of Special Interest by System Organ Class and Preferred Term (Safety Population)3 |
| Table 14.3-2.1.1 – Summary of Hematology Laboratory Data (Safety Population) |
| Table 14.3-2.1.2 – Outside of Normal Range - Shift Table for Hematology Laboratory Parameters (Safety Population) |
| Table 14.3-2.1.3 – Clinician Assessment - Shift Table for Hematology Laboratory Parameters (Safety Population) |
| Table 14.3-2.1.4 – On-study Hematology Adverse Events: Worst NCI-CTCAE Grade per patient (Safety Population) |
| Table 14.3-2.1.5 – Shift table of Worst NCI-CTCAE Grade for Hematological parameters (Safety Population)4 |



(TFL shells):

| Table 14.3-2.2.1 – Summary of Clinical Chemistry Laboratory Data (Safety Population) | 42 |
|---|---|
| Table 14.3-2.2.2 – Outside of Normal Range - Shift Table for Clinical Chemistry Laboratory Parameters (Safety Population) | 42 |
| Table 14.3-2.2.3 – Clinician Assessment - Shift Table for Clinical Chemistry Laboratory Parameters (Safety Population) | 42 |
| Table 14.3-2.2.4 – On-study Clinical Chemistry Adverse Events: Worst NCI-CTCAE Grade per patient (Safety Population) | 42 |
| Table 14.3-2.2.5 – Shift table of Worst NCI-CTCAE Grade for Clinical Chemistry Laboratory parameters (Safety Population) | 43 |
| Table 14.3-2.3.1 – Summary of Coagulation Laboratory Data (Safety Population) | 43 |
| Table 14.3-2.4 – Summary of Thyroid Panel Laboratory Data (Safety Population) | 43 |
| Table 14.3-2.5.1 – Summary of Urinalysis Laboratory Data (Safety Population) | 44 |
| Table 14.3-2.5.2 – Outside of Normal Range - Shift Table for Urinalysis Laboratory Parameters (Safety Population) | 44 |
| Table 14.3-2.5.3 – Clinician Assessment - Shift Table for Urinalysis Laboratory Parameters (Safety Population) | 44 |
| Table 14.3-2.5.4 – On-study Urinalysis Adverse Events: Worst NCI-CTCAE Grade per patient (Safety Population) | 44 |
| Table 14.3-2.5.5 – Shift table of Worst NCI-CTCAE Grade for Urinalysis Laboratory parameters (Safety Population) | 45 |
| Table 14.3-2.6 – Summary of Other Laboratory Data (Safety Population) | 46 |
| Table 14.3-3.1 – Summary of Vital Signs (Safety Population) | 47 |



(TFL shells):

| Table 14.3-3.2 – Summary of Abnormal Vital Signs (Safety Population) | 48 |
|---|---|
| Table 14.3-4.1 – Summary of ECG Parameters (Safety Population) | 51 |
| Table 14.3-4.2 – Summary of Abnormal ECG Intervals (Safety Population) | 52 |
| Listing 16.1.7-1 – Treatment Administration (All Patients) | 54 |
| Listing 16.1.7-2 – Infusion Interruption (All Patients) | 55 |
| Listing 16.2.1-1.1 – Preface to Inclusion and Exclusion Criteria | 56 |
| Listing 16.2.1-1.2 – List of Failed Inclusion and Exclusion Criteria (All Patients) | 57 |
| Listing 16.2.1-2 – Patient Disposition (All Patients) | 58 |
| Listing 16.2.2 – Protocol Deviations (All Patients) | 59 |
| Listing 16.2.3-1 – Demographic and Baseline Characteristics (All Patients) | 60 |
| Listing 16.2.3-2 – HIV, Hepatitis and Pregnancy Test Results (All Patients) | 61 |
| Listing 16.2.4-1 – Cancer History (All Patients) | 63 |
| Listing 16.2.4-2 – Prior Cancer Therapies (All Patients) | 64 |
| Listing 16.2.4-3 – Other Medical History (All Patients) | 65 |



(TFL shells):

| Listing 16.2.4-4 – Cardiac Function (All Patients) | 66 |
|---|---|
| Listing 16.2.4-5 – Ophthalmologic Exam (All Patients) | 67 |
| Listing 16.2.4-6 – RECIST Target Lesions (All Patients) | 68 |
| Listing 16.2.4-7 – RECIST Non-Target Lesions (All Patients) | 69 |
| Listing 16.2.4-8 – Prior and Concomitant Medications (All Patients) | 70 |
| Listing 16.2.5 – Drug Exposure (All Patients) | 71 |
| Listing 16.2.6-1 – Urine concentrations of CPX-POM and Metabolites (All Patients) | 72 |
| Listing 16.2.6-2 – Plasma concentrations of CPX-POM and Metabolites (All Patients) | 72 |
| Listing 16.2.6-3 – Plasma concentrations of Biomarkers Assays (All Patients) | 73 |
| Listing 16.2.6-4 – PBMC Biomarkers Assays (All Patients) | 73 |
| Listing 16.2.6-5 – Urine beta-glucuronidase activity (All Patients) | 74 |
| Listing 16.2.7-1 – Adverse Events (All Patients) | 75 |
| Listing 16.2.7-2 – Serious Adverse Events (All Patients) | 76 |
| Listing 16.2.7-3 – Adverse Events Leading to Discontinuation (All Patients) | 76 |



(TFL shells):

| Listing 16.2.7-4 – Adverse Events Leading to Death (All Patients) | 76 |
|---|---|
| Listing 16.2.8-1 – Patients Laboratory Profile: Hematology (All Patients) | 77 |
| Listing 16.2.8-2 – Patients Laboratory Profile: Clinical Chemistry (All Patients) | 78 |
| Listing 16.2.8-3 – Patients Laboratory Profile: Coagulation and Thyroid Panel (All Patients) | 78 |
| Listing 16.2.8-4 – Patients Laboratory Profile: Urinalysis (All Patients) | 78 |
| Listing 16.2.8-5 – Vital Signs (All Patients) | 79 |
| Listing 16.2.8-6 – ECG Results and Interpretation (All Patients) | 80 |



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE --- Page 1 of Y

## Table 14.1-1 - Patients disposition (All patients)

| Cycle | CPX-POM<br>30 mg/m^2<br>N=1<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM [D3] mg/m^2 N=X n (%) | CPX-POM [D4] mg/m^2 N=X n (%) | CPX-POM [D5] mg/m^2 N=X n (%) | CPX-POM<br>[D6] mg/m^2<br>N=X<br>n (%) | CPX-POM<br>[D7] mg/m^2<br>N=X<br>n (%) |
|---|---|---|---|---|---|---|---|
| Cycle 1 | | | | | | | |
| Treated | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Completed the cycle [a] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Discontinued from the cycle | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Reason for discontinuation from the cycle | | | | | | | |
| Dose Limitimg Toxicity | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Withdrawn Consent | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Physician Decision | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Death | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lost to Follow-up | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Percentages are based on the number of patients enrolled.

[a] A patient completed Cycle 1 if s/he attended visit Day 10 (if Cycle 1 was not the last cycle) or Visit Day 22 (if Cycle 1 was the last cycle).

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 2 of Y

# Table 14.1-1 - Patients disposition (All patients)

| Cycle | CPX-POM<br>30 mg/m^2<br>N=1<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM [D3] mg/m^2 N=X n (%) | CPX-POM<br>[D4] mg/m^2<br>N=X<br>n (%) | CPX-POM [D5] mg/m^2 N=X n (%) | CPX-POM [D6] mg/m^2 N=X n (%) | CPX-POM<br>[D7] mg/m^2<br>N=X<br>n (%) |
|---|---|---|---|---|---|---|---|
| Cycle 2 | | | | | | | |
| Treated | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Completed the cycle [b] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Discontinued from the cycle | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Reason for discontinuation from the cycle | | | | | | | |
| Dose Limitimg Toxicity | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Withdrawn Consent | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Physician Decision | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Death | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lost to Follow-up | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

#### <repeat until last-1 cycle>

Percentages are based on the number of patients enrolled.

[b] A patient completed Cycle 2 (or any next cycle until last-1 cycle) if s/he attended visit Day 6 (if Cycle 2 or any next cycle was not the last cycle) or Visit Day 22 (if Cycle 2 or any next cycle was the last cycle).

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)



Sponsor: CicloMed
Protocol: CPX-POM-001

Statistical Analysis Plan

(TFL shells):


Filename: (Specify file name.rtf)

Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page X of Y

### Table 14.1-1 - Patients disposition (All patients enrolled)

| Cycle | CPX-POM<br>30 mg/m^2<br>N=1<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM [D3] mg/m^2 N=X n (%) | CPX-POM [D4] mg/m^2 N=X n (%) | CPX-POM [D5] mg/m^2 N=X n (%) | CPX-POM [D6] mg/m^2 N=X n (%) | CPX-POM [D7] mg/m^2 N=X n (%) |
|---|---|---|---|---|---|---|---|
| Last Cycle | | | | | | | |
| Treated | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Completed the cycle [c] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Discontinued from the cycle | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Reason for discontinuation from the cycle | | | | | | | |
| Dose Limitimg Toxicity | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Withdrawn Consent | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Physician Decision | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Death | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lost to Follow-up | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Attended the follow-up visit (Day 28) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Percentages are based on the number of patients enrolled.

[c] A patient completed the Last Cycle if s/he attended visit Day 22.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

#### PROGRAMMING NOTES:

• Display all the reasons for discontinuation where there is at least one patient within that category



**Sponsor**: CicloMed

Protocol: CPX-POM-001 Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- 

Table 14.1-2 - Number (%) of Patients in the Analysis Populations (All patients)

| | CPX-POM<br>30 mg/m^2<br>N=1<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM [D3] mg/m^2 N=X n (%) | CPX-POM [D4] mg/m^2 N=X n (%) | CPX-POM [D5] mg/m^2 N=X n (%) | CPX-POM<br>[D6] mg/m^2<br>N=X<br>n (%) | CPX-POM<br>[D7] mg/m^2<br>N=X<br>n (%) |
|---|---|---|---|---|---|---|---|
| Safety Population | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Efficacy Population | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| PK Population | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Percentages are based on the number of enrolled patients.

The Safety population includes all patients who have received at least one dose of CPX-POM.

The Efficacy population includes all patients who have received at least one dose of CPX-POM, had RECIST measurable disease at baseline and had at least one other post-baseline tumor assessment.

The PK population includes all patients for whom at least one plasma and/or urine sample has been obtained and analyzed for determination of plasma drug and metabolites concentration.

Program: (Program name.sas) (run on: DDMMYYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

• For the safety population, patients are displayed based on the actually received treatment.



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- 

Table 14.1-3 - Summary of Demography (ITT Population)

| | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM |
|---|---|---|---|---|---|---|---|
| | 30 mg/m^2 | [D2] mg/m^2 | [D3] mg/m^2 | [D4] mg/m^2 | [D5] mg/m^2 | [D6] mg/m^2 | [D7] mg/m^2 |
| | N=1 | N=X | N=X | N=X | N=X | N=X | N=X |
| Age [a] (years) | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |
| Age group [n (%)] | | | | | | | |
| < 65 years | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ≥ 65 years | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Sex [n (%)] | | | | | | | |
| Male | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Female | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Race [n (%)] | | | | | | | |
| White | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Black or African American | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Asian | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| American Indian or Alaska Native | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Native Hawaiian or | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other Pacific Islander<br>Other | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

<sup>[</sup>a] Age at Screening.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

<sup>[</sup>b] Body mass index (BMI)  $(kg/m^2)$  = Weight (kg) /  $(Height (m))^2$ .

<sup>[</sup>c] The denominator is the number of females in each dose group.



(TFL shells):



(TFL shells):


Filename: (Specify file name.rtf)

Protocol: CPX-POM-001 --- DELIVERY TYPE ---- 

Table 14.1-3 - Summary of Demography (ITT Population)

| | CPX-POM<br>30 mg/m^2<br>N=1 | CPX-POM<br>[D2] mg/m^2<br>N=X | CPX-POM<br>[D3] mg/m^2<br>N=X | CPX-POM [D4] mg/m^2 N=X | CPX-POM<br>[D5] mg/m^2<br>N=X | CPX-POM<br>[D6] mg/m^2<br>N=X | CPX-POM [D7] mg/m^2 N=X |
|---|---|---|---|---|---|---|---|
| Female of child bearing potential | | | | | | | |
| [n (%)] [c] | | | | | | | |
| Yes | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| No | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Country [n (%)] | | | | | | | |
| XXXXX | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| XXXXX | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| XXXXX | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Height (cm) | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |

<sup>[</sup>a] Age at Screening.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

<sup>[</sup>b] Body mass index (BMI)  $(kg/m^2)$  = Weight (kg) / (Height (m))\*\*2.

<sup>[</sup>c] The denominator is the number of females in each dose group.



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---

Table 14.1-3 - Summary of Demography (ITT Population)

| | CPX-POM<br>30 mg/m^2 | CPX-POM<br>[D2] mg/m^2 | CPX-POM<br>[D3] mg/m^2 | CPX-POM [D4] mg/m^2 | CPX-POM<br>[D5] mg/m^2 | CPX-POM [D6] mg/m^2 | CPX-POM<br>[D7] mg/m^2 |
|---|---|---|---|---|---|---|---|
| | N=1 | N=X | N=X | N=X | N=X | N=X | N=X |
| Weight (kg) | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |
| BMI [b] (kg/m^2) | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |
| BSA [d] (kgxm) | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |

<sup>[</sup>a] Age at Screening.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)


<sup>[</sup>b] Body Mass Index (BMI)  $(kg/m^2) = Weight (kg) / (Height (m))^2$ .

<sup>[</sup>c] The denominator is the number of females in each dose group.

<sup>[</sup>d] Body Surface Area (BSA)  $(kgxm) = 0.007184 \times Weight (kg)^0.425 / (Height (m))^0.725 (Dubois formula).$ 



(TFL shells):



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

### Table 14.1-4 - Protocol Deviations (Safety Population)

| Protocol Deviations Category | CPX-POM<br>30 mg/m^2<br>N=1<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM [D3] mg/m^2 N=X n (%) | CPX-POM<br>[D4] mg/m^2<br>N=X<br>n (%) | CPX-POM [D5] mg/m^2 N=X n (%) | CPX-POM [D6] mg/m^2 N=X n (%) | CPX-POM [D7] mg/m^2 N=X n (%) |
|---|---|---|---|---|---|---|---|
| Any Protocol Deviations | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| <pre>Inclusion / Exclusion Criteria INCL01 <cont.></cont.></pre> | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Prohibited Medications | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) |

### <cont.>

A patient could be counted under more than one category.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

• Categories are from the protocol deviations criteria form, the table only shows examples.



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- 

# Table 14.1-5.1 - Disease Characteristics (Safety Population)

| | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM |
|---|---|---|---|---|---|---|---|
| | 30 mg/m^2 | [D2] mg/m^2 | [D3] mg/m^2 | [D4] mg/m^2 | [D5] mg/m^2 | [D6] mg/m^2 | [D7] mg/m^2 |
| | N=1 | N=X | N=X | N=X | N=X | N=X | N=X |
| Cancer Type? [n (%)] | | | | | | | |
| Solid Tumor | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lymphoma | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Solid Tumor Organ Site [n (%)] | | | | | | | |
| Lung | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Breast | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Colon | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Prostate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Time since first diagnosis of Cance | r (months) | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |
| Disease Stage at the Cancer diagnos | is date? [n | (%)] | | | | | |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Disease Stage at Screening visit da | te? [n (%)] | | | | | | |
| 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |




(TFL shells):


Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Protocol: CPX-POM-001

--- DELIVERY TYPE ----

Filename: (Specify file name.rtf)


Table 14.1-5.1 - Disease Characteristics (Safety Population)

| | | (201200] | , roparacrom, | | | | |
|---|---|---|---|---|---|---|---|
| | CPX-POM<br>30 mg/m^2<br>N=1 | CPX-POM<br>[D2] mg/m^2<br>N=X | CPX-POM<br>[D3] mg/m^2<br>N=X | CPX-POM [D4] mg/m^2 N=X | CPX-POM<br>[D5] mg/m^2<br>N=X | CPX-POM<br>[D6] mg/m^2<br>N=X | CPX-POM<br>[D7] mg/m^2<br>N=X |
| Presence of metastases? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Time between date of Metastatic of | diagnosis and d | ate of Cycle 1 | visit Day 1 | (months) | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |
| Extent of current Metastatic dise | ease | | | | | | |
| Bone? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lungs? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Liver? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Pelvic Lymph Nodes? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Extrapelvic Lymph Nodes? [n (%) | 1 | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other? [n (%)] | , , , | , , | , , | , , | , , | | , |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 110 | 2121 (2121 • 21) | 7777 (7777 • 77) | 1111 (1111 • 11) | 1111 (1111 • 11) | 1111 (1111 • 11) | (2323 * 23 / | (2121 • 21) |




(TFL shells):


Yes XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X)

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Table 14.1-5.2 - Other Medical History (Safety Population)

| System Organ Class/<br>Preferred Term | CPX-POM<br>30 mg/m^2<br>N=1<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM [D3] mg/m^2 N=X n (%) | CPX-POM [D4] mg/m^2 N=X n (%) | CPX-POM [D5] mg/m^2 N=X n (%) | CPX-POM [D6] mg/m^2 N=X n (%) | CPX-POM [D7] mg/m^2 N=X n (%) |
|---|---|---|---|---|---|---|---|
| At least one other previous condition? | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| System Organ Class #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <etc></etc> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System Organ Class #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <etc></etc> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

#### PROGRAMMING NOTES:

• The Primary System Organ Classes are presented by alphabetical order and the Preferred Terms are sorted within Primary System Organ Classes by alphabetical order.

Filename: (Specify file name.rtf)



(TFL shells):



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Table 14.1-6.1.1 - Prior Medications by Therapeutic Class and Preferred Term (Safety Population)

| Therapeutic Class/<br>Preferred Term | CPX-POM<br>30 mg/m^2<br>N=1<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM [D3] mg/m^2 N=X n (%) | CPX-POM [D4] mg/m^2 N=X n (%) | CPX-POM [D5] mg/m^2 N=X n (%) | CPX-POM [D6] mg/m^2 N=X n (%) | CPX-POM [D7] mg/m^2 N=X n (%) |
|---|---|---|---|---|---|---|---|
| At least one prior medication? | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Therapeutic Class #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <etc></etc> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Therapeutic Class #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <etc></etc> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

A prior medication is a medication whose end date is before the date of first CPX-POM dose.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

#### PROGRAMMING NOTES:

• The Therapeutic Classes are presented by alphabetical order and the Preferred Terms are sorted within Therapeutic Classes by alphabetical order.

Filename: (Specify file name.rtf)

• A medication / therapy can appear within more than one Therapeutic Class.



(TFL shells):


Table 14.1-6.1.2 - Concomitant Medications by Therapeutic Class and Preferred Term (Safety Population)

#### Replicate of Table 14.1-6.1.1

#### PROGRAMMING NOTES:

- Update foootnote: replace 'A prior medication is a medication whose end date is before the date of first CPX-POM dose' by 'A concomitant medication is a medication that started before the date of first dose and stopped on (or is ongoing after) the date of first dose OR a medication whose start date is either the same as (or after) the date of first dose'.
- Update 'At least one prior medication' by 'At least one concomitant medication'.
- The Therapeutic Classes are presented by alphabetical order and the Preferred Terms are sorted within Therapeutic Classes by alphabetical order.
- A medication / therapy can appear within more than one Therapeutic Class.



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE --- 

Table 14.1-7 - Overall Exposure to Study Drug and Drug Compliance (Safety Population)

| | CPX-POM<br>30 mg/m^2<br>N=1 | CPX-POM [D2] mg/m^2 N=X | CPX-POM [D3] mg/m^2 N=X | CPX-POM [D4] mg/m^2 N=X | CPX-POM [D5] mg/m^2 N=X | CPX-POM<br>[D6] mg/m^2<br>N=X | CPX-POM<br>[D7] mg/m^2<br>N=X |
|---|---|---|---|---|---|---|---|
| Study Drug Exposure (days) [a] | | | | | | | |
| beauf brag Emposaro (aufo, [u] | XX | XX | XX | XX | XX | XX | XX |
| n | | | | | | | |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |
| Study Drug Exposure (mg) [b] | | | | | | | |
| | XX | XX | XX | XX | XX | XX | XX |
| n | | | | | | | |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |

<sup>[</sup>a] The CPX-POM exposure expressed in days is defined as the number of days between the first dose taken date and the last dose taken date + 1 day.

Filename: (Specify file name.rtf)

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

<sup>[</sup>b] The CPX-POM exposure expressed in mg is defined as: dose per m^2 x Body Surface Area x CPX-POM exposure expressed in days.



**Sponsor**: CicloMed

Protocol: CPX-POM-001
Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- 

Table 14.2.1 - Patients who have had at least one other post-baseline tumor assessment (Efficacy Population)

| | CPX-POM<br>30 mg/m^2<br>N=1 | CPX-POM [D2] mg/m^2 N=X | CPX-POM<br>[D3] mg/m^2<br>N=X | CPX-POM<br>[D4] mg/m^2<br>N=X | CPX-POM [D5] mg/m^2 N=X | CPX-POM<br>[D6] mg/m^2<br>N=X | CPX-POM<br>[D7] mg/m^2<br>N=X |
|---|---|---|---|---|---|---|---|
| At least one other post-baseline tumor assessment | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Primary Tumor Site [n (%)] | | | | | | | |
| Primary Tumor Site #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Primary Tumor Site #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Primary Tumor Site #3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <etc></etc> | | | | | | | |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

• A last column with the header 'CPX-POM All Doses' will also be displayed.



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- 

## Table 14.2.2 - Summary of Patients Responses (Efficacy Population)

| Visit/ | CPX-POM<br>30 mg/m^2 | CPX-POM [D2] mg/m^2 | CPX-POM [D3] mg/m^2 | CPX-POM [D4] mg/m^2 | CPX-POM<br>[D5] mg/m^2 | CPX-POM [D6] mg/m^2 | CPX-POM [D7] mg/m^2 |
|---|---|---|---|---|---|---|---|
| Type of Response | N=1 | N=X | N=X | N=X | N=X | N=X | N=X |
| Cycle 2-Day 1 Visit | | | | | | | |
| Target Lesion Response [n (%)] | | | | | | | |
| Complete Response | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Partial Response | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Stable Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not evaluable | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Non-Target Lesion Response [n ( | %)] | | | | | | |
| Complete Response | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Partial Response | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Stable Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not evaluable | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Overall Response [n (%)] | | | | | | | |
| Complete Response | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Partial Response | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Stable Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive Disease | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not evaluable | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

<repeat for Day 1 visit of each cycle from Cycle 3 to last Cycle number over all patients>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

• A last column with the header 'CPX-POM All Doses' will also be displayed.



(TFL shells):



Sponsor: CicloMed
Protocol: CPX-POM-001

Statistical Analysis Plan

Filename: (Specify file name.rtf)

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- 

Table 14.3-1.1 - Overview of Adverse Events (Safety Population)

| | CPX-POM<br>30 mg/m^2<br>N=1<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM<br>[D3] mg/m^2<br>N=X<br>n (%) | CPX-POM<br>[D4] mg/m^2<br>N=X<br>n (%) | CPX-POM [D5] mg/m^2 N=X n (%) | CPX-POM [D6] mg/m^2 N=X n (%) | CPX-POM<br>[D7] mg/m^2<br>N=X<br>n (%) |
|---|---|---|---|---|---|---|---|
| Number of patients with | | | | | | | |
| at least one: | | | | | | | |
| AE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| TEAE * | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Related TEAE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| TEAE leading to discontinuation | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Related TEAE leading to | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| discontinuation | | | | | | | |
| Serious TEAE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Serious related TEAE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

<sup>\*</sup> A treatment-emergent adverse events (TEAE) is defined as an adverse event which started on or after the first dose of CPX-POM administration.

MedDRA version <version number>.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

#### PROGRAMMING NOTES:

- "Leading to discontinuation" is derived from action taken = permanently discontinued.
- A last column with the header 'CPX-POM All Doses' will also be displayed.



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Table 14.3-1.2 - Number (%) of Patients with Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population)

| System Organ Class/<br>Preferred Term | CPX-POM<br>30 mg/m^2<br>N=1<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM [D3] mg/m^2 N=X n (%) | CPX-POM [D4] mg/m^2 N=X n (%) | CPX-POM [D5] mg/m^2 N=X n (%) | CPX-POM [D6] mg/m^2 N=X n (%) | CPX-POM [D7] mg/m^2 N=X n (%) |
|---|---|---|---|---|---|---|---|
| Number of patients with at least one TEAE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System Organ Class #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #3 <etc></etc> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| \e\c\/ | | | | | | | |
| System Organ Class #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #3 <etc></etc> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

If there was more than one TEAE reported under the same System Organ Class and Preferred Term, the patient was counted only once under that System Organ Class and that Preferred Term. If there was more than one TEAE reported under the same System Organ Class, the patient was counted only once under that System Organ Class.

MedDRA version <version number>.

Filename: (Specify file name.rtf)

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

#### PROGRAMMING NOTES:

• The System Organ Classes are presented by decreasing frequency (within the total column - all CPX-POM doses groups combined - not displayed) and the Preferred Terms within a System Organ Class are presented by decreasing frequency (within the total column - all CPX-POM doses groups combined - not displayed).



(TFL shells):


Table 14.3-1.3 - Number (%) of Patients with Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population)

#### Replicate of Table 14.3-1.2

Table 14.3-1.4 - Number (%) of Patients with Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population)

#### Replicate of Table 14.3-1.2

Table 14.3-1.5 - Number (%) of Patients with Serious Related Treatment-Emergent Adverse Events by System Organ Class and
Preferred Term
(Safety Population)

#### Replicate of Table 14.3-1.2

Table 14.3-1.6 - Number (%) of Patients with Treatment-Emergent Adverse Events Leading to Discontinuation by System Organ Class and Preferred Term (Safety Population)

#### Replicate of Table 14.3-1.2

#### PROGRAMMING NOTES:

• "Leading to discontinuation" is derived from action taken = permanently discontinued.



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Table 14.3-1.7 - Number (%) of Patients with Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Maximal Severity (Safety Population)

| System Organ Class/ Preferred Term/ Maximal severity | CPX-POM<br>30 mg/m^2<br>N=1<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM<br>[D3] mg/m^2<br>N=X<br>n (%) | CPX-POM [D4] mg/m^2 N=X n (%) | CPX-POM [D5] mg/m^2 N=X n (%) | CPX-POM<br>[D6] mg/m^2<br>N=X<br>n (%) | CPX-POM [D7] mg/m^2 N=X n (%) |
|---|---|---|---|---|---|---|---|
| Number of patients with any TEAE | | | | | | | |
| Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System Organ Class #1 | | | | | | | |
| Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #1 | | | | | | | |
| Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

If there was more than one TEAE reported under the same System Organ Class and Preferred Term, the patient was counted only once under the maximal severity for that System Organ Class and Preferred Term. If there was more than one TEAE reported under the same System Organ Class, the patient was counted only once under the maximal severity for that System Organ Class.

MedDRA version System Organ Class

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

#### PROGRAMMING NOTES:

- Display all severities even if there are no patients.
- The System Organ Classes are presented by decreasing frequency (within the total column all CPX-POM doses groups combined not displayed) and the Preferred Terms within a System Organ Class are presented by decreasing frequency (within the

Filename: (Specify file name.rtf)



(TFL shells):


total column - all CPX-POM doses groups combined - not displayed).

Table 14.3-1.8 - Number (%) of Patients with Related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Maximum Severity (Safety Population)

Replicate of Table 14.3-1.7



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Table 14.3-1.9 - Number (%) of Patients with Treatment-Emergent Adverse Events of Special Interest by System Organ Class and
Preferred Term
(Safety Population)

| System Organ Class/ | CPX-POM<br>30 mg/m^2<br>N=1 | CPX-POM<br>[D2] mg/m^2<br>N=X | CPX-POM [D3] mg/m^2 N=X | CPX-POM [D4] mg/m^2 N=X | CPX-POM<br>[D5] mg/m^2<br>N=X | CPX-POM<br>[D6] mg/m^2<br>N=X | CPX-POM<br>[D7] mg/m^2<br>N=X |
|---|---|---|---|---|---|---|---|
| Preferred Term | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Number of patients with at least one TEAE of Special Interest | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System Organ Class #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <etc></etc> | | | | | | | |
| System Organ Class #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term #3 <etc></etc> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

The TEAEs of Special Interest are the clinically significant ophthalmological abnormalities.

If there was more than one TEAE of Special Interest reported under the same System Organ Class and Preferred Term, the patient was counted only once under that System Organ Class and that Preferred Term. If there was more than one TEAE of Special Interest reported under the same System Organ Class, the patient was counted only once under that System Organ Class.

MedDRA version <version number>.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

#### PROGRAMMING NOTES:

• The System Organ Classes are presented by decreasing frequency for all CPX-POM doses groups combined and the Preferred Terms within a System Organ Class are presented by decreasing frequency for all CPX-POM doses groups combined.

Filename: (Specify file name.rtf)

• A last column with the header 'CPX-POM All Doses' will also be displayed.



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Table 14.3-2.1.1 - Summary of Hematology Laboratory Data (Safety Population)

Laboratory Parameter: Hemoglobin (unit)

| | CPX-POM | | CPX-POM [D3] mg/m^2 N=X | CPX-POM<br>[D4] mg/m^2 | CPX-POM | CPX-POM | CPX-POM<br>[D7] mg/m^2<br>N=X |
|---|---|---|---|---|---|---|---|
| | 30 mg/m^2 | | | | [D5] mg/m^2 | [D6] mg/m^2 | |
| | N=1 | N=X | | N=X | N=X | N=X | |
| Baseline [a] | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |
| Cycle 1-Day 4 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |
| Change from Baseline | | | | | | | |
| to Cycle 1-Day 4 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX |

<repeat for Cycle 1 Day 10 visit>

<for Cycle 2 to last-1 Cycle, repeat for Day 1 visit and Day 4 visit>
<for the last Cycle, repeat for Day 22 visit and Day 28 follow-up visit>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

<sup>[</sup>a] Baseline was the last value/result of assessment prior to or on day of first study treatment.



(TFL shells):


#### PROGRAMMING NOTES:

Repeat for all hematology parameters: Hemoglobin, Hematocrit, Platelet count, RBC count, Reticulocytes, WBC Count with Differential, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils.
 Protocol: CPX-POM-001

Table 14.3-2.1.2 - Outside of Normal Range - Shift Table for Hematology Laboratory Parameters (Safety Population)

Dose group : CPX-POM 30 mg/m^2 (N=1)

| | | | Baseline [a] value | | | |
|---|---|---|---|---|---|---|
| Parameter/ | Value | Low | Normal | High | Low/High* | |
| Visit | at Visit | n (%) | n (%) | n (%) | n (%) | Total |
| Hemoglobin (unit) | | | | | | |
| Cycle 1-Day 4 (N**=XX) | Low | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Normal | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | High | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Low/High* | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Total | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX |
| Cycle 1-Day 10 (N**=XX) | Low | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Normal | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | High | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Low/High* | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Total | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX |

<for Cycle 2 to last-1 Cycle, repeat for Day 1 visit and Day 4 visit>
<for the last Cycle, repeat for Day 22 visit and Day 28 follow-up visit>
<repeat for all doses groups>

Percentage was based on the number of patients present at each visit with non-missing results for the considered parameter.

\* Included patients with Low or High results. \*\* Denominator of the percentage.

[a] Baseline was the last value/result of assessment prior to or on day of first study treatment intake.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

#### PROGRAMMING NOTES:

• Repeat for all doses groups.

Filename: (Specify file name.rtf)


(TFL shells):


• Repeat for all hematology parameters: Hemoglobin, Hematocrit, Platelet count, RBC count, Reticulocytes, WBC Count with Differential, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils.



Sponsor: CicloMed
Protocol: CPX-POM-001

Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Table 14.3-2.1.3 - Clinician Assessment - Shift Table for Hematology Laboratory Parameters (Safety Population)

Dose group : CPX-POM 30 mg/m^2 (N=1)

| | Baseline [a] value | | | | |
|---|---|---|---|---|---|
| Parameter/ | Value | Normal | Abnormal, NCS | Abnormal, CS | |
| Visit | at Visit | n (%) | n (%) | n (%) | Total |
| Hemoglobin (unit) | | | | | |
| Cycle 1-Day 4 (N*=XX) | Normal | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Abnormal, NCS | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Abnormal, CS | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Total | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX |
| Cycle 1-Day 10 (N*=XX) | Normal | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Abnormal, NCS | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Abnormal, CS | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Total | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX |

<for Cycle 2 to last-1 Cycle, repeat for Day 1 visit and Day 4 visit> <for the last Cycle, repeat for Day 22 visit and Day 28 follow-up visit> <repeat for the other hematology parameters>

<repeat for all doses groups>

Percentage was based on the number of patients present at each visit with non-missing results for the considered parameter.

\* Denominator of the percentage.

[a] Baseline was the last value/result of assessment prior to or on day of first study treatment. CS = Clinically Significant; NCS = Not Clinically Significant.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

## Filename: (Specify file name.rtf)

- Repeat for all doses groups.
- Repeat for all hematology parameters: Hemoglobin, Hematocrit, Platelet count, RBC count, Reticulocytes, WBC Count with Differential, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils.



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Table 14.3-2.1.4 - On-study Hematology Adverse Events: Worst NCI-CTCAE Grade per patient (Safety Population)

| Parameter/<br>Worst NCI-CTCAE grade | CPX-POM<br>30 mg/m^2<br>N=1<br>n (%) | CPX-POM [D2] mg/m^2 N=X n (%) | CPX-POM [D3] mg/m^2 N=X n (%) | CPX-POM [D4] mg/m^2 N=X n (%) | CPX-POM<br>[D5] mg/m^2<br>N=X<br>n (%) | CPX-POM<br>[D6] mg/m^2<br>N=X<br>n (%) | CPX-POM [D7] mg/m^2 N=X n (%) |
|---|---|---|---|---|---|---|---|
| Hemoglobin (unit) | | | | | | | |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Grade 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Grade 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Grade 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Grade 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Hematocrit (unit) | | | | | | | |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Grade 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Grade 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Grade 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Grade 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

#### <repeat for the other hematology parameters>

For a given laboratory parameter, a patient must have at least one on-study grade assessed to be included.

For a given laboratory parameter, the number of treated patients with at least one on-study grade assessed for that parameter will be used as the denominator for the calculation of percentages.

A patient with multiple results for a parameter will only be counted under the maximum NCI-CTCAE grade for this parameter. Laboratory ranges are based on NCI-CTCAE version 4.0.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

## PROGRAMMING NOTES:

• Repeat for all hematology parameters: Hemoglobin, Hematocrit, Platelet count, RBC count, Reticulocytes, WBC Count with

Filename: (Specify file name.rtf)



(TFL shells):


Differential, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils.



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Table 14.3-2.1.5 - Shift table of Worst NCI-CTCAE Grade for Hematological parameters (Safety Population)

| | | | | | Worst NCI-C | TCAE grade | | |
|---|---|---|---|---|---|---|---|---|
| | Baseline | Normal | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Missing | Total |
| Parameter | grade | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (응) |
| Hematocrit (unit) | Normal | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Grade 1 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Grade 2 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Grade 3 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Grade 4 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Missing | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Total | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | _ | | | | | | | |
| Hemoglobin (unit) | Normal | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Grade 1 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Grade 2 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Grade 3 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Grade 4 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Missing | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| | Total | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |

#### <repeat for the other hematology parameters>

For a given laboratory parameter, a patient must have at least one baseline and one on-treatment grades assessed to be included. For a given laboratory parameter, the number of treated patients with at least one baseline and one on-treatment grades assessed for that parameter will be used as the denominator for the calculation of percentages.

A patient with multiple results for a parameter will only be counted under the maximum NCI-CTCAE grade for this parameter. Laboratory ranges are based on NCI-CTCAE version 4.0.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

# PROGRAMMING NOTES:

• Repeat for all hematology parameters: Hemoglobin, Hematocrit, Platelet count, RBC count, Reticulocytes, WBC Count with Differential, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils.

Filename: (Specify file name.rtf)



(TFL shells):


Table 14.3-2.2.1 - Summary of Clinical Chemistry Laboratory Data (Safety Population)

#### Replicate of Table 14.3-2.1.1

#### PROGRAMMING NOTES:

Clinical Chemistry parameters are: Potassium, Sodium, Chloride, Glucose, BUN, Creatinine, Creatinine clearance, ALP, ALT, AST, GGT, Alkaline phosphatase, Direct bilirubin, Indirect bilirubin, Total bilirubin, Total protein, Albumin, Calcium, Bicarbonate, Magnesium, Phosphate, Lipase, Amylase

Table 14.3-2.2.2 - Outside of Normal Range - Shift Table for Clinical Chemistry Laboratory Parameters (Safety Population)

#### Replicate of Table 14.3-2.1.2

#### PROGRAMMING NOTES:

Clinical Chemistry parameters are: Potassium, Sodium, Chloride, Glucose, BUN, Creatinine, Creatinine clearance, ALP, ALT, AST, GGT, Alkaline phosphatase, Direct bilirubin, Indirect bilirubin, Total bilirubin, Total protein, Albumin, Calcium, Bicarbonate, Magnesium, Phosphate, Lipase, Amylase

Table 14.3-2.2.3 - Clinician Assessment - Shift Table for Clinical Chemistry Laboratory Parameters (Safety Population)

#### Replicate of Table 14.3-2.1.3

#### PROGRAMMING NOTES:

Clinical Chemistry parameters are: Potassium, Sodium, Chloride, Glucose, BUN, Creatinine, Creatinine clearance, ALP, ALT, AST, GGT, Alkaline phosphatase, Direct bilirubin, Indirect bilirubin, Total bilirubin, Total protein, Albumin, Calcium, Bicarbonate, Magnesium, Phosphate, Lipase, Amylase

Table 14.3-2.2.4 - On-study Clinical Chemistry Adverse Events: Worst NCI-CTCAE Grade per patient (Safety Population)

#### Replicate of Table 14.3-2.1.4

#### PROGRAMMING NOTES:

Clinical Chemistry parameters are: Potassium, Sodium, Chloride, Glucose, BUN, Creatinine, Creatinine clearance, ALP, ALT, AST,




GGT, Alkaline phosphatase, Direct bilirubin, Indirect bilirubin, Total bilirubin, Total protein, Albumin, Calcium, Bicarbonate, Magnesium, Phosphate, Lipase, Amylase

Table 14.3-2.2.5 - Shift table of Worst NCI-CTCAE Grade for Clinical Chemistry Laboratory parameters (Safety Population)

#### Replicate of Table 14.3-2.1.5

#### PROGRAMMING NOTES:

Clinical Chemistry parameters are: Potassium, Sodium, Chloride, Glucose, BUN, Creatinine, Creatinine clearance, ALP, ALT, AST, GGT, Alkaline phosphatase, Direct bilirubin, Indirect bilirubin, Total bilirubin, Total protein, Albumin, Calcium, Bicarbonate, Magnesium, Phosphate, Lipase, Amylase

Table 14.3-2.3.1 - Summary of Coagulation Laboratory Data (Safety Population)

### Replicate of Table 14.3-2.1.1

#### PROGRAMMING NOTES:

- Coagulation parameters are PT and aPTT.
- Only Day 1 visit of each cycle

Table 14.3-2.4 - Summary of Thyroid Panel Laboratory Data (Safety Population)

### Replicate of Table 14.3-2.1.1

- Coagulation parameters are TSH, Free T4 and Free and total T3
- Only Day 1 visit of each cycle



(TFL shells):


Table 14.3-2.5.1 - Summary of Urinalysis Laboratory Data (Safety Population)

#### Replicate of Table 14.3-2.1.1

#### PROGRAMMING NOTES:

- Urinalysis parameters are Color, Turbidity, pH, Specific gravity, Glucose, Ketones, Nitrites, Bilirubin, Urobilirubin, Protein, RBCs, WBCs, Epithelial cells, Casts, Crystals, Bacteria, eGFR (Screening only)
- Replace 'Day 4' by 'Day 5' for each cycle

Table 14.3-2.5.2 - Outside of Normal Range - Shift Table for Urinalysis Laboratory Parameters (Safety Population)

#### Replicate of Table 14.3-2.1.2

#### PROGRAMMING NOTES:

- Urinalysis parameters are Color, Turbidity, pH, Specific gravity, Glucose, Ketones, Nitrites, Bilirubin, Urobilirubin, Protein, RBCs, WBCs, Epithelial cells, Casts, Crystals, Bacteria, eGFR (Screening only)
- Replace 'Day 4' by 'Day 5' for each cycle

Table 14.3-2.5.3 - Clinician Assessment - Shift Table for Urinalysis Laboratory Parameters (Safety Population)

#### Replicate of Table 14.3-2.1.3

#### PROGRAMMING NOTES:

- Urinalysis parameters are Color, Turbidity, pH, Specific gravity, Glucose, Ketones, Nitrites, Bilirubin, Urobilirubin, Protein, RBCs, WBCs, Epithelial cells, Casts, Crystals, Bacteria, eGFR (Screening only)
- Replace 'Day 4' by 'Day 5' for each cycle

Table 14.3-2.5.4 - On-study Urinalysis Adverse Events: Worst NCI-CTCAE Grade per patient (Safety Population)

Replicate of Table 14.3-2.1.4




(TFL shells):


#### PROGRAMMING NOTES:

• Urinalysis parameters are Color, Turbidity, pH, Specific gravity, Glucose, Ketones, Nitrites, Bilirubin, Urobilirubin, Protein, RBCs, WBCs, Epithelial cells, Casts, Crystals, Bacteria, eGFR (Screening only)

• Replace 'Day 4' by 'Day 5' for each cycle

Table 14.3-2.5.5 - Shift table of Worst NCI-CTCAE Grade for Urinalysis Laboratory parameters (Safety Population)

Replicate of Table 14.3-2.1.5

- Urinalysis parameters are Color, Turbidity, pH, Specific gravity, Glucose, Ketones, Nitrites, Bilirubin, Urobilirubin, Protein, RBCs, WBCs, Epithelial cells, Casts, Crystals, Bacteria, eGFR (Screening only)
- Replace 'Day 4' by 'Day 5' for each cycle



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ----

### Table 14.3-2.6 - Summary of Other Laboratory Data (Safety Population)

| | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM |
|---|---|---|---|---|---|---|---|
| Visit/ | 30 mg/m^2 | [D2] mg/m^2 | [D3] mg/m^2 | | [D5] mg/m^2 | [D6] mg/m^2 | [D7] mg/m^2 |
| Parameter | N=1 | N=X | N=X | N=X | N=X | N=X | N=X |
| Screening visit | | | | | | | |
| HIV? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Hepatitis A? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Hepatitis B? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Hepatitis C? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Pregnancy test? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Cycle 1-Day 1 | | | | | | | |
| Pregnancy test? [n (%)] | | | | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)



(TFL shells):


Table 14.3-3.1 - Summary of Vital Signs (Safety Population)

Replicate of Table 14.3-2.1.1

- Update "laboratory parameter" by "parameter"
- Vital signs include pulse rate, blood pressure, respiratory rate, oxygen saturation and temperature
- On Days 1 and 5, vital signs are measured at pre-dose and at 6-hour intervals post-dose.



Protocol: CPX-POM-001
Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- 

# Table 14.3-3.2 - Summary of Abnormal Vital Signs (Safety Population)

| Parameter/ | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM |
|---|---|---|---|---|---|---|---|
| Visit/ | 30 mg/m^2 | [D2] mg/m^2 | [D3] mg/m^2 | [D4] mg/m^2 | [D5] mg/m^2 | [D6] mg/m^2 | [D7] mg/m^2 |
| Category | N=1 | N=X | N=X | N=X | N=X | N=X | N=X |
| Pulse rate (bpm) | | | | | | | |
| Cycle 1 | | | | | | | |
| Baseline [a]* | XX | XX | XX | XX | XX | XX | XX |
| > 150 bpm | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| [101-150] bpm | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| < 55 bpm | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Cycle 1-Day 2 * | XX | XX | XX | XX | XX | XX | XX |
| > 150 bpm | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| [101-150] bpm | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| < 55 bpm | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |

<repeat for next Cycle 1 visits>

<for Cycle 2 to last-1 Cycle, repeat for Day 1 visit to Day 6 visit>

<for the last Cycle, repeat for Day 1 visit to Day 6 visit, Day 22 visit and Day 28 follow-up visit>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

<sup>\*</sup> Denominator for the percentages.

<sup>[</sup>a] Baseline was the last value/result of assessment prior to or on day of first study treatment.

<sup>&</sup>gt; 150 bpm: Very High values [101-150] bpm: High values

<sup>&</sup>lt; 55 bpm: Low values



Sponsor: CicloMed
Protocol: CPX-POM-001

Statistical Analysis Plan

Filename: (Specify file name.rtf)

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- 

# Table 14.3-3.2 - Summary of Abnormal Vital Signs (Safety Population)

| Parameter/ | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM |
|---|---|---|---|---|---|---|---|
| Visit/ | 30 mg/m^2 | [D2] mg/m^2 | [D3] mg/m^2 | [D4] mg/m^2 | [D5] mg/m^2 | [D6] mg/m^2 | [D7] mg/m^2 |
| Category | N=1 | N=X | N=X | N=X | N=X | N=X | N=X |
| Systolic Blood Pressure (mmHg) | | | | | | | |
| Baseline [a]* | XX | XX | XX | XX | XX | XX | XX |
| >= 161 mmHg | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| [131-160] bpm | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| < 95 mmHg | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Cycle 1-Day 2 * | XX | XX | XX | XX | XX | XX | XX |
| >= 161 mmHg | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| [131-160] bpm | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| < 95 mmHg | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |

#### <repeat for next Cycle 1 visits>

<for Cycle 2 to last-1 Cycle, repeat for Day 1 visit to Day 6 visit>
<for the last Cycle, repeat for Day 1 visit to Day 6 visit, Day 22 visit and Day 28 follow-up visit>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

<sup>\*</sup> Denominator for the percentages.

<sup>[</sup>a] Baseline was the last value/result of assessment prior to or on day of first study treatment.

<sup>&</sup>gt;= 161 bpm: Very High values

<sup>[131-160]</sup> bpm: High values

<sup>&</sup>lt; 95 bpm: Low values



Sponsor: CicloMed
Protocol: CPX-POM-001

Statistical Analysis Plan

Filename: (Specify file name.rtf)

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- 

Table 14.3-3.2 - Summary of Abnormal Vital Signs (Safety Population)

| Parameter/ | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM |
|---|---|---|---|---|---|---|---|
| Visit/ | 30 mg/m^2 | [D2] mg/m^2 | [D3] mg/m^2 | [D4] mg/m^2 | [D5] mg/m^2 | [D6] mg/m^2 | [D7] mg/m^2 |
| Category | N=1 | N=X | N=X | N=X | N=X | N=X | N=X |
| Diastolic Blood Pressure (mmHg) | | | | | | | |
| Baseline [a]* | XX | XX | XX | XX | XX | XX | XX |
| >= 101 mmHg | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| [86-100] bpm | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| < 50 mmHg | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Cycle 1-Day 2 * | XX | XX | XX | XX | XX | XX | XX |
| >= 101 mmHg | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| [86-100] bpm | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| < 50 mmHg | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |

#### <repeat for next Cycle 1 visits>

<for Cycle 2 to last-1 Cycle, repeat for Day 1 visit to Day 6 visit>
<for the last Cycle, repeat for Day 1 visit to Day 6 visit, Day 22 visit and Day 28 follow-up visit>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

<sup>\*</sup> Denominator for the percentages.

<sup>[</sup>a] Baseline was the last value/result of assessment prior to or on day of first study treatment.

<sup>&</sup>gt;= 101 bpm: Very High values [86-100] bpm: High values

<sup>&</sup>lt; 50 bpm: Low values



(TFL shells):


Table 14.3-4.1 - Summary of ECG Parameters (Safety Population)

Replicate of Table 14.3-2.1.1

- Update "laboratory parameter" by "ECG parameter"
- Include all ECG parameters



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of Y

Table 14.3-4.2 - Summary of Abnormal ECG Intervals (Safety Population)

| Parameter/ | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM | CPX-POM |
|---|---|---|---|---|---|---|---|
| Visit/ | 30 mg/m^2 | [D2] mg/m^2 | [D3] mg/m^2 | [D4] mg/m^2 | [D5] mg/m^2 | [D6] mg/m^2 | [D7] mg/m^2 |
| Category | N=1 | N=X | N=X | N=X | N=X | N=X | N=X |
| Heart rate (bpm) | | | | | | | |
| Baseline [a]* | XX | XX | XX | XX | XX | XX | XX |
| Normal | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Abnormal, NCS | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Abnormal, CS | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Cycle 1-Day 5 * | XX | XX | XX | XX | XX | XX | XX |
| Normal | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Abnormal, NCS | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Abnormal, CS | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |

<for Cycle 2 to last-1 cycle, repeat for Day 1 visit>
<for last cycle, repeat for Day 1 visit and Day 28 follow-up visit>
<repeat for PR interval and QRS interval>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

<sup>\*</sup> Denominator for the percentages.

<sup>[</sup>a] Baseline was the last value/result of assessment prior to or on day of first study treatment. CS = Clinically Significant; NCS = Not Clinically Significant.



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page X of Y

# Table 14.3-4.2 - Summary of Abnormal ECG Intervals (Safety Population)

| Parameter/<br>Visit/<br>Category | CPX-POM<br>30 mg/m^2<br>N=1 | CPX-POM [D2] mg/m^2 N=X | CPX-POM [D3] mg/m^2 N=X | CPX-POM [D4] mg/m^2 N=X | CPX-POM<br>[D5] mg/m^2<br>N=X | CPX-POM [D6] mg/m^2 N=X | CPX-POM [D7] mg/m^2 N=X |
|---|---|---|---|---|---|---|---|
| QTcB interval (msec) | | | | | | | |
| Baseline [a]* | XX | XX | XX | XX | XX | XX | XX |
| > 450 msec | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| > 480 msec | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| > 500 msec | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Cycle 1-Day 5 * | XX | XX | XX | XX | XX | XX | XX |
| > 450 msec | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| > 480 msec | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| > 500 msec | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Change from Baseline to Cycle 1-Day 5 * | XX | XX | XX | XX | XX | XX | XX |
| > 30 msec | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| > 60 msec | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |

<for Cycle 2 to last-1 cycle, repeat for Day 1 visit>
<for last cycle, repeat for Day 28 follow-up visit>
<repeat for QTcF interval>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

PROGRAMMING NOTES: For QTcF interval, the category '> 500 msec' will be replaced by '> 500 msec (CS)' and the category '> 60 msec' will be replaced by '> 60 msec (CS)'.

<sup>\*</sup> Denominator for the percentages.

<sup>[</sup>a] Baseline was the last value/result of assessment prior to or on day of first study treatment. CS = Clinically Significant; NCS = Not Clinically Significant.



**Sponsor**: CicloMed **Protocol**: CPX-POM-001

Statistical Analysis Plan (TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE --- Page 1 of X

Listing 16.1.7-1 - Treatment Administration (All Patients)

| Center/<br>Patient | Visit | CPX-POM<br>Dose group | CPX-POM<br>Dose<br>Amount<br>per<br>Prot.? | If no, Reason for Adjustment? | Total Inf. Bag vol. of Sal. and CPX-POM (ml) | Was<br>Total<br>Vol.<br>Inf.? | If no, actual Vol. Inf.? | Adm. Date (Day) Inf. Start Time- Inf. End Time | Arm<br>Used<br>for IV | Infusion<br>Interrupted? |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXXXX | BAS | 30 mg/m^2 | Yes | | XXX | Yes | | DDMMMYYYY (XX) | Right | |
| | C1 TRT D2 | 30 mg/m^2 | Yes | | Yes | Yes | | HH:MM-HH:MM DDMMMYYYY (XX) | Right | |
| | C1 TRT D3 | 30 mg/m^2 | Yes | | XXX | Yes | | HH:MM-HH:MM DDMMMYYYY (XX) | Right | |
| | C1 TRT D4 | 30 mg/m^2 | Yes | | XXX | Yes | | HH:MM-HH:MM DDMMMYYYY (XX) | Right | |
| | C1 TRT D5 | 30 mg/m^2 | No | Adverse event | XXX | No | XXX | HH:MM-HH:MM DDMMMYYYY (XX) HH:MM-HH:MM | Right | Yes [a] |

#### <repeat for Days 1,2,3,4 and 5 of next cycles if relevant>

Prot.: Protocol; Inf.: Infusion/Infused; Vol.: Volume; Sal.: Saline; Adm.: Administration; Inter.: Interruption/Interrupted;

IV: Intravenous

[a]: see further details regarding the infusion interruption in Listing 16.1.7-2

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:



Protocol: CPX-POM-001
Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ----


Listing 16.1.7-2 - Infusion Interruption (All Patients)

| Center/<br>Patient | Visit | CPX-POM<br>Dose group | Reason for Inf. Inter.? | Specify | Adm. Date (Day)<br>Time Inf. Inter. | Inf.<br>Rest.? | Time Inf.<br>Restarted | Reason<br>for Not<br>Restarting? | Specify | Inf.<br>Site<br>React.? |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXXXX | C1 TRT D5 | 30 mg/m^2 | Infusion reaction | XXXXX | DDMMMYYYY (XX)<br>HH:MM | No | | Infusion reaction | XXXXX | Yes |
| XXXXXXX | C2 TRT D2 | [D2] mg/m^2 | Technical problem | XXXXX | DDMMMYYYY (XX)<br>HH:MM | Yes | нн:мм | | XXXXX | No |

#### <cont>

Inf.: Infusion; Inter.: Interrupted; Rest.: Restarted; React.: Reaction.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Listing 16.2.1-1.1 - Preface to Inclusion and Exclusion Criteria

| Protocol<br>Version | Inclusion/<br>Exclusion No. | Inclusion / Exclusion Text |
|---|---|---|
| 3.0 | INCL01 | Patient has histologically- or cytologically- confirmed metastatic or advanced-stage solid malignant tumor that is refractory to standard therapy. Patients should only be included if no therapy exists or if they have received all standard therapies that would be potentially curative or might provide significant benefit. |
| | INCL02 | Patient may have received up to 4 prior lines of cytotoxic chemotherapy or immunotherapy for their metastatic disease (e.g., docetaxel + doxorubicin ± cyclophosphamide), and also may have received additional prior endocrine therapy, as appropriate (e.g., for breast or prostate cancer), or non-myelosuppressive therapy (e.g., bevacizumab, trastuzumab). |
| | <etc></etc> | |
| | EXCL01 | Patient has a history of risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome) or requires the use of concomitant medications that prolong the QT/QTc interval during study participation. |
| | EXCL02 | Patient has an abnormal cardiac appearance/heart size, as evidenced by chest X-ray or computed tomography (CT) scan. |
| | <etc></etc> | |

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

- List all Inclusion / Exclusion criteria as per eCRF.
- Note: Inclusion / Exclusion text displayed in the listing shell is based on the text in Protocol Version 3.0.



Protocol: CPX-POM-001
Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ----

Listing 16.2.1-1.2 - List of Failed Inclusion and Exclusion Criteria


Filename: (Specify file name.rtf)

| Center/<br>Patient | CPX-POM<br>Dose group | Protocol<br>Version | Failed Inclusion / Exclusion |
|---|---|---|---|
| XXXX | [D3] mg/m^2 | 3.0 | INCL01, INCL09 EXCL05, EXCL08, EXC110 |
| XXXX | [D5] mg/m^2 | 3.0 | INCL02<br>EXCL03, EXCL07 |

(All Patients)

<to be completed with the other patients having at least one protocol deviation>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

- List all Inclusion / Exclusion criteria that are failed (i.e. 'N' for inclusion and 'Y' for exclusion)
- Listing to be sorted by increasing CPX-POM dose.



Sponsor: CicloMed
Protocol: CPX-POM-001

Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ----


# Listing 16.2.1-2 - Patient Disposition (All Patients)

| Center/ | | CPX-POM | Date (day) of Discontinuation/ | Reason for | Date (day) of | Date (day) of | |
|---|---|---|---|---|---|---|---|
| Patient | Country | Dose group | Completion | Discontinuation | Last Dose | Death | Reason |
| XXXX | XXX | 30 mg/m^2 | DDMMMYYYY (XXX) | | DDMMMYYYY (XXX) | | |
| XXXX | XXX | [D2] mg/m^2 | DDMMMYYYY (XXX) | | DDMMMYYYY (XXX) | | |
| XXXX | XXX | [D3] mg/m^2 | DDMMMYYYY (XXX) | | DDMMMYYYY (XXX) | | |
| XXXX | XXX | [D4] mg/m^2 | DDMMMYYYY (XXX) | | DDMMMYYYY (XXX) | | |
| XXXX | XXX | [D4] mg/m^2 | DDMMMYYYY (XXX) | Adverse Event | DDMMMYYYY (XXX) | | |
| XXXX | XXX | [D4] mg/m^2 | DDMMMYYYY (XXX) | | DDMMMYYYY (XXX) | | |

#### <etc>

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Listing 16.2.2 - Protocol Deviations (All Patients)

| | | | | Leading to Exclusion | |
|---|---|---|---|---|---|
| Center/ | CPX-POM | | | from Analysis | Analysis |
| Patient | Dose group | Category | Details | Population? | Population(s) |
| XXXX | [D4] mg/m^2 | Compliance | Not treated | Yes | SAFETY |

### <to be completed with the other patients having at least one protocol deviation>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:



Protocol: CPX-POM-001
Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Listing 16.2.3-1 - Demographic and Baseline Characteristics (All Patients)

| Center/<br>Patient | Country | CPX-POM<br>Dose group | Date of<br>Birth | Age<br>(year) | Sex | Race | Weight<br>(kg) | Height<br>(cm) | BMI<br>(kg/m^2) | BSA<br>(kgxm) | Patient of Child Bearing Potential? | Creat.<br>Clear.<br>(unit) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | XXX | 30 mg/m^2 | DDMMMYYYY | XX | Male | XXXXX | XXX.X | XXX | XX.X | XX.X | | XXX |
| XXXX | XXX | [D2] mg/m^2 | DDMMMYYYY | XX | Female | XXXXX | XXX.X | XXX | XX.X | XX.X | Yes | XXX |
| XXXX | XXX | [D3] mg/m^2 | DDMMMYYYY | XX | Female | XXXXX | XXX.X | XXX | XX.X | XX.X | No | XXX |
| XXXX | XXX | [D4] mg/m^2 | DDMMMYYYY | XX | Male | XXXXX | XXX.X | XXX | XX.X | XX.X | | XXX |
| XXXX | XXX | [D4] mg/m^2 | DDMMMYYYY | XX | Male | XXXXX | XXX.X | XXX | XX.X | XX.X | | XXX |
| XXXX | XXX | [D4] mg/m^2 | DDMMMYYYY | XX | Female | XXXXX | XXX.X | XXX | XX.X | XX.X | No | XXX |

#### <etc>

Creat. Clear.: Creatinine Clearance.

Dates are displayed as DDMMMYYYY, -- represents an unknown date component. Age was calculated from date of birth and date of screening. BMI  $(kg/m^2)$  = Weight (kg) /(Height (m)^2. BSA (kgxm) = 0.007184 x Weight (kg)^0.425 / (Height (m))^0.725 (Dubois formula).

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:



Sponsor: CicloMed Protocol: CPX-POM-001

Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Listing 16.2.3-2 - HIV, Hepatitis and Pregnancy Test Results (All Patients)

| Center/<br>Patient | CPX-POM<br>Dose group | Visit | Parameter | Assessment Performed? | Assessment<br>Date | Study<br>Day | Result |
|---|---|---|---|---|---|---|---|
| XXXX | 30 mg/m^2 | SCR | HIV | Yes | DDMMMYYYY | XX | No |
| | - | | Hepatitis A | Yes | DDMMMYYYY | XX | No |
| | | | Hepatitis B | Yes | DDMMMYYYY | XX | No |
| | | | Hepatitis C | Yes | DDMMMYYYY | XX | No |
| | | | Pregnancy Test | Yes | DDMMMYYYY | XX | No |
| | | BAS | Pregnancy Test | Yes | DDMMMYYYY | XX | No |

<repeat for Day 1 of next cycles if relevant>
<cont.>

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:



(TFL shells):




(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Listing 16.2.4-1 - Cancer History (All Patients)

| Center/<br>Patient | CPX-POM<br>Dose group | Cancer<br>Type | If Other, specify | Initial<br>Diagnosis<br>Date (Day) | Disease<br>Stage at<br>Initial<br>Diagnosis | Current<br>Disease<br>Stage | Pres.<br>of<br>Metas.? | Date of<br>Metastatic<br>Diagnosis (Day) | Location | If Other, specify |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | 30 mg/m^2 | XXXXX | | DDMMMYYYY (XXX) | Grade X | Grade X | No | | | |
| XXXX | [D2] mg/m^2 | XXXXX | | DDMMMYYYY (XXX) | Grade X | Grade X | No | | | |
| XXXX | [D3] mg/m^2 | XXXXX | | DDMMMYYYY (XXX) | Grade X | Grade X | Yes | DDMMMYYYY (XXX) | Bone | |
| XXXX | [D4] mg/m^2 | XXXXX | | YYYY | Grade X | Grade X | No | | | |
| XXXX | [D4] mg/m^2 | Other | XXXXX | DDMMMYYYY (XXX) | Grade X | Grade X | Yes | DDMMMYYYY (XXX) | Other | XXXXX |
| XXXX | [D4] mg/m^2 | XXXXX | | | Grade X | Grade X | Yes | DDMMMYYYY (XXX) | Lungs<br>Liver | |

#### <etc>

Pres.: Presence; Metas.: Mestastases

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:



Protocol: CPX-POM-001 Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE --- Page 1 of X

Listing 16.2.4-2 - Prior Cancer Therapies (All Patients)

| Center/<br>Patient | CPX-POM<br>Dose group | Therapy<br>Type | If Radiation, specify | Therapy<br>Name | Line of<br>Therapy | Treatment<br>Setting | Treatment<br>Intent | Start Date (Day)<br>End Date (Day) | Best<br>Response |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | 30 mg/m^2 | XXXXX | | XXXXX | X | XXXXX | XXXXX | DDMMMYYYY (XX)<br>DDMMMYYYY (XX) | XXXXX |
| XXXX | [D2] mg/m^2 | XXXXX | | XXXXX | X | XXXXX | XXXXX | DDMMMYYYY (XX)<br>DDMMMYYYY (XX) | XXXXX |
| XXXX | [D3] mg/m^2 | Radiation | XXXXX | XXXXX | X | XXXXX | XXXXX | DDMMMYYYY (XX) | XXXXX |
| (ata) | | | | | | | | DDMMMYYYY (XX) | |

#### <etc>

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:



Protocol: CPX-POM-001
Statistical Analysis Plan

Filename: (Specify file name.rtf)

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Listing 16.2.4-3 - Other Medical History (All Patients)

CPX-POM Dose Group: 30 mg/m^2

| Center/<br>Patient | System Organ Class/<br>Preferred Term/<br>Verbatim | Start Date (Day) | End Date (Day) | Treated with medication? |
|---|---|---|---|---|
| XXXX | XXXXXX/<br>XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (XXX) | DDMMMYYYY (XXX) | No |
| XXXX | XXXXXX/<br>XXXXXX/<br>XXXXXXXXXX | MMMYYYY | Ongoing | Yes |

#### <cont.>

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

MedDRA <version no.>

PROGRAMMING NOTES:

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)



Protocol: CPX-POM-001
Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Listing 16.2.4-4 - Cardiac Function (All Patients)

| Center/<br>Patient | CPX-POM<br>Dose group | Echocardiogram or MUGA Scan performed? | Method of<br>Assessment | Date of<br>Assessment | Overall<br>Interpretation | If Abnormal CS, specify |
|---|---|---|---|---|---|---|
| XXXX | 30 mg/m^2 | Yes | Echocardiogram | DDMMMYYYY | XXXXX | |
| XXXX | [D2] mg/m^2<br>[D3] mg/m^2 | Yes<br>Yes | MUGA<br>Echocardiogram | DDMMMYYYY<br>DDMMMYYYY | Abnormal CS<br>XXXXX | XXXXX |
| <etc></etc> | _ | | - | | | |

CS: Clinically Significant. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:



Protocol: CPX-POM-001
Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Listing 16.2.4-5 - Ophthalmologic Exam (All Patients)

| Center/<br>Patient | CPX-POM<br>Dose group | Ophthalmology<br>Assessments<br>performed? | Use of<br>Corrective<br>Lenses? | Date of<br>Assessment | Overall<br>Interpretation | If Abnormal CS, specify |
|---|---|---|---|---|---|---|
| XXXX | 30 mg/m^2 | Yes | Yes | DDMMMYYYY | XXXXX | |
| XXXX | [D2] mg/m^2 | Yes | No | DDMMMYYYY | Abnormal CS | XXXXX |
| XXXX | [D3] mg/m^2 | Yes | No | DDMMMYYYY | XXXXX | |
| <etc></etc> | | | | | | |

CS: Clinically Significant. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:



Protocol: CPX-POM-001
Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

# Listing 16.2.4-6 - RECIST Target Lesions (All Patients)

| Center/<br>Patient | CPX-POM<br>Dose group | Visit/<br>Target Lesions<br>Identified at<br>Screening Visit? | Date of<br>Scans<br>review | Lesion<br>Number | Organ<br>Site | Specific<br>Location<br>within the<br>Organ Site | Lymph<br>Node<br>Type | Method | Lesion<br>Diameter<br>(mm) |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | 30 mg/m^2 | C1 TRT D1 / Yes | DDMMMYYYY | T01 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| | | | | T02 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| XXXX | [D2] mg/m^2 | C1 TRT D1 / Yes | DDMMMYYYY | T01 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| | | C2 TRT D1 / Yes | DDMMMYYYY | T01 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| | | | DDMMMYYYY | T02 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| XXXX | [D2] mg/m^2 | C1 TRT D1 / Yes | DDMMMYYYY | T01 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| | | C2 TRT D1 / Yes | DDMMMYYYY | T01 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| | | C3 TRT D1 / Yes | DDMMMYYYY | T01 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |

#### <etc>

CS: Clinically Significant. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:



Protocol: CPX-POM-001
Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

# Listing 16.2.4-7 - RECIST Non-Target Lesions (All Patients)

| Center/<br>Patient | CPX-POM<br>Dose group | Visit/<br>Non-Target<br>Lesions<br>Identified at<br>Screening Visit? | Date of<br>Scans<br>review | Lesion<br>Number | Organ<br>Site | Specific<br>Location<br>within the<br>Organ Site | Lymph<br>Node<br>Type | Method | Result |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | 30 mg/m^2 | C1 TRT D1 / Yes | DDMMMYYYY | NT01 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| | | | | NT02 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| XXXX | [D2] mg/m^2 | C1 TRT D1 / Yes | DDMMMYYYY | NT01 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| | | C2 TRT D1 / Yes | DDMMMYYYY | NT01 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| | | | | NT02 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| | | | | NT03 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| XXXX | [D2] mg/m^2 | C1 TRT D1 / Yes | DDMMMYYYY | NT01 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| | - | C2 TRT D1 / Yes | DDMMMYYYY | NT01 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| | | C3 TRT D1 / Yes | DDMMMYYYY | NT01 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |

#### <etc>

CS: Clinically Significant. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

# Listing 16.2.4-8 - Prior and Concomitant Medications (All Patients)

CPX-POM Dose Group: 30 mg/m^2

| Center/<br>Patient | Type of<br>Medication | Therapeutic Class<br>Preferred Term<br>Verbatim | Start Date (Day)/<br>End Date (Day) | Total Daily Dose<br>(unit)/<br>Frequency/<br>Route | Reason/<br>Indication |
|---|---|---|---|---|---|
| XXXX | | XXXXXX/<br>XXXXXX/<br>XXXXXXXXXXX | DDMMMYYYY (<-180)/<br>DDMMMYYYY (XXX) | XXXXXXXX (XXX)/ Once/ Inhalation | xxxxxxxxxxx |
| | Conc.** Proh. [a] | XXXXXX/<br>XXXXXXXXXXXXXXX | MMMYYYY/<br>Ongoing | Other, XXXX/<br>bid/<br>Cutaneous | XXXXXX |
| XXXX | Prior* | XXXXXX/<br>XXXXXX/<br>XXXXXXXXXX | MMMYYYY/<br>DDMMMYYYY (XXX) | 200 mg/<br>tid/<br>Other, XXXXX | xxxxxxxxxxxxxxx |

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

[a] Proh. = Prohibited medication.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

#### PROGRAMMING NOTES:

- Listing to be sorted by increasing CPX-POM dose.
- Use abbreviations or codes to present data if not enough space (and add appropriate abbreviations / codes in footnotes).

Filename: (Specify file name.rtf)

<sup>\*</sup> Prior = any medication whose end date is before the date of first dose.

<sup>\*\*</sup> Conc. = any medication that started before the date of first dose and stopped on (or is ongoing after) the date of first dose OR any medication whose start date is either the same as (or after) the date of first dose.



Protocol: CPX-POM-001
Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Listing 16.2.5 - Drug Exposure (All Patients)

| Center/<br>Patient | CPX-POM<br>Dose group | Date of first dose admnistration | Visit of<br>last dose<br>admnistration | Date of last dose admnistration | Exposure<br>(days) | Exposure (mg) |
|---|---|---|---|---|---|---|
| XXXX | 30 mg/m^2 | DDMMMYYYY | C1 TRT D5 | DDMMMYYYY | XX | XX |
| XXXX | [D2] mg/m^2 | DDMMMYYYY | C2 TRT D5 | DDMMMYYYY | XX | XX |

#### <cont.>

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY.

The CPX-POM exposure expressed in days is defined as the number of days between the first dose taken date and the last dose taken date + 1 day.

The CPX-POM exposure expressed in mg is defined as: dose per m<sup>2</sup> x Body Surface Area x CPX-POM exposure expressed in days.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:



Protocol: CPX-POM-001
Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Listing 16.2.6-1 - Urine concentrations of CPX-POM and Metabolites (All Patients)

CPX-POM Dose Group: 30 mg/m^2

| Center/<br>Patient | Parameter<br>(Unit) | Visit | Assessment Sample | Assess | ment<br>Time | Study<br>Day | Urine<br>Volume<br>(mL) | CPX-POM<br>Conc.<br>(ng/mL) | CPX<br>Conc.<br>(ng/mL) | CPX-G<br>Conc.<br>(ng/mL) |
|---|---|---|---|---|---|---|---|---|---|---|
| | CPX-POM | | | | | | | | | |
| XXXX | (XXXX) | C1 TRT D1 | Pre-Dose | DDMMMYYYY | HH:MM | | XX | XX | XX | XX |
| | | | Post-Dose [0-12] | DDMMMYYYY | HH:MM | | XX | XX | XX | XX |
| | | | Post-Dose [12-24] | DDMMMYYYY | HH:MM | | XX | XX | XX | XX |
| | | C1 TRT D5 | Post-Dose [0-12] | DDMMMYYYY | HH:MM | XX | XX | XX | XX | XX |
| | | | Post-Dose [12-24] | DDMMMYYYY | HH:MM | XX | XX | XX | XX | XX |

Conc.: Concentration.

Study Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component. Baseline was the last non-missing assessment prior or on the first dose date. SI units and results presented. ND = Not Done.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

•

Listing 16.2.6-2 - Plasma concentrations of CPX-POM and Metabolites (All Patients)

Replicate of Listing 16.2.6-1



Sponsor: CicloMed
Protocol: CPX-POM-001

Statistical Analysis Plan (TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Listing 16.2.6-3 - Plasma concentrations of Biomarkers Assays (All Patients)

CPX-POM Dose Group: 30 mg/m^2

| Center/<br>Patient | Parameter<br>(Unit) | Visit | Assessment<br>Sample | Assessi | ment<br>Time | Study<br>Day | VEGF<br>Conc.<br>(pg/mL) | Percent<br>change<br>from<br>Baseline | IL-6<br>Conc.<br>(pg/mL) | change<br>from<br>Baseline | IL-8<br>Conc.<br>(pg/mL) | change<br>from<br>Baseline |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | CPX-POM(XXXX) | C1 TRT D1<br>C1 TRT D5 | Pre-Dose<br>Pre-Dose | DDMMMYYYY<br>DDMMMYYYY | | XX | XX<br>XX | XX.X | XX<br>XX | XX.X | XX<br>XX | XX.X |

# <repeat for Day 1 and Day 5 visits of next cycles if relevant> <repeat for Day 22 visit of last cycle>

Conc.: Concentration.

The Baseline concentrations are the concentrations obtained at Day 1 Visit of Cycle 1.

Study Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component. Baseline was the last non-missing assessment prior or on the first dose date. SI units and results presented.

ND = Not Done.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

• Repeat for all doses groups.

Listing 16.2.6-4 - PBMC Biomarkers Assays (All Patients)

#### Replicate of Listing 16.2.6-3

- PBMC Biomarkers are Notch 1, surviving, cyclin D, c-Myc and Hes 1 using RT-PCR.
- Repeat for all doses groups.



Protocol: CPX-POM-001
Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Listing 16.2.6-5 - Urine beta-glucuronidase activity (All Patients)

CPX-POM Dose Group: 30 mg/m^2

| Center/<br>Patient | Parameter (Unit) | Visit | Assessment Sample | Assessi | ment<br>Time | Study<br>Day | Urine beta-glucuronidase activity (U/mL) |
|---|---|---|---|---|---|---|---|
| XXXX | CPX-POM (XXXX) | C1 TRT D1 | Post-Dose [0-12]<br>Post-Dose [12-24] | DDMMMYYYY<br>DDMMMYYYY | | | XX<br>XX |
| | | C1 TRT D5 | Post-Dose [0-12]<br>Post-Dose [12-24] | DDMMMYYYY<br>DDMMMYYYY | | XX<br>XX | XX<br>XX |

Study Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component. Baseline was the last non-missing assessment prior or on the first dose date. SI units and results presented. ND = Not Done.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

• Repeat for all doses groups.



Protocol: CPX-POM-001
Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Listing 16.2.7-1 - Adverse Events (All Patients)

CPX-POM Dose Group: 30 mg/m^2

| Center/<br>Patient | System Organ Class/<br>Preferred Term/<br>Verbatim | Start Date (Day)/<br>End Date (Day) | Action Taken/<br>Medication or<br>Therapies Taken? | Outcome/<br>Severity/<br>Relationship | SAE? |
|---|---|---|---|---|---|
| XXXX | XXXXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXXXXXX | DDMMMYYYY (XXX)/<br>DDMMMYYYY (XXX) | None/<br>No | XXXXXXX/<br>Mild/<br>Not related | No |
| | XXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (XXX)/<br>Ongoing | Dose Adjusted/<br>Yes | Resolved/<br>Moderate/<br>Definitely related | Yes |
| XXXX | XXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXX/<br>XXXXXX | DDMMMYYYY (XXX)/<br>MMMYYYY | | XXXXXXXX/<br>XXXXXX/<br>XXXXXXX | No |

#### <cont.>

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component.

Filename: (Specify file name.rtf)

MedDRA version <version #>.

PROGRAMMING NOTES:

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

• Repeat for the other CPX-POM doses by increasing order.



(TFL shells):


Listing 16.2.7-2 - Serious Adverse Events (All Patients)

### Replicate of Listing 16.2.7-1

#### PROGRAMMING NOTES:

- Repeat for the other CPX-POM doses by increasing order.
- Select all AEs where SAE = Yes.
- Remove column 'SAE' and remove SAE from footnote.

Listing 16.2.7-3 - Adverse Events Leading to Discontinuation (All Patients)

#### Replicate of Listing 16.2.7-1

#### PROGRAMMING NOTES:

- Repeat for the other CPX-POM doses by increasing order.
- Select all AEs where action taken = permanently discontinued.

Listing 16.2.7-4 - Adverse Events Leading to Death (All Patients)

### Replicate of Listing 16.2.7-1

- Repeat for the other CPX-POM doses by increasing order.
- Select all AEs where outcome = Fatal



Protocol: CPX-POM-001 Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Listing 16.2.8-1 - Patients Laboratory Profile: Hematology (All Patients)

CPX-POM Dose Group: 30 mg/m^2

| Center/ | | Assess | ment | Study | Parameter | <u>-</u> | Normal | | | CTCAE | Change<br>from | Clinical |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient | Visit | Date | Time | Day | (Unit) | | Range | Res | ult | grade | Baseline | Interpretation |
| XXXX | BAS | DDMMMYYYY | HH:MM | XXX | XXXXXXXX | (XXXX) | XXXXXX | XX | | Grade 1 | | Normal |
| | C1 TRT D1 | DDMMMYYYY | HH:MM | XXX | XXXXXXXX | (XXXX) | XXXXXX | XX | L/H | Grade 2 | XXXX | Abnormal, NCS |
| | C1 TRT D4 | DDMMMYYYY | HH:MM | XXX | XXXXXXXX | (XXXX) | XXXXXX | XX | L/H | Grade 2 | XXXX | Abnormal, NCS |
| | C1 TRT D10 | DDMMMYYYY | HH:MM | XXX | XXXXXXXX | (XXXX) | XXXXXX | XX | L/H | Grade 3 | XXXX | Abnormal, CS |

<for Cycle 2 to last-1 cycle, repeat for Day 1 visit and Day 4 visit if relevant> <for the last cycle, repeat also for Day 22 visit and Day 28 visit>

Study Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY, -- represents an unknown date component. Baseline was the last non-missing assessment prior or on the first dose date. SI units and results presented. L/H = low/high value based upon normal ranges. R = repeat/unscheduled assessments. CS = Clinically Significant; NCS = Not Clinically Significant; ND = Not Done.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

Repeat for the other CPX-POM doses by increasing order.



(TFL shells):


Listing 16.2.8-2 - Patients Laboratory Profile: Clinical Chemistry (All Patients)

#### Replicate of Listing 16.2.8-1

#### PROGRAMMING NOTES:

• Listing to be sorted by increasing order.

Listing 16.2.8-3 - Patients Laboratory Profile: Coagulation and Thyroid Panel (All Patients)

### Replicate of Listing 16.2.8-1

#### PROGRAMMING NOTES:

- Listing to be sorted by increasing order.
- Only Day 1 of each cycle.

Listing 16.2.8-4 - Patients Laboratory Profile: Urinalysis (All Patients)

#### Replicate of Listing 16.2.8-1

- Listing to be sorted by increasing order.
- Replace 'Day 4' by 'Day 5' for each cycle.



(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Listing 16.2.8-5 - Vital Signs (All Patients)

CPX-POM Dose Group: 30 mg/m^2

| Center/<br>Patient | Visit | Assessment<br>Date Time | Study<br>Day | Parameter (unit) | Position | Result | Change from<br>Baseline |
|---|---|---|---|---|---|---|---|
| XXXX | BAS | DDMMMYYYY HH:MM | XXX | Pulse Rate (bpm) Respiratory Rate (bpm) Systolic BP (mmHg) Diastolic BP (mmHg) Oxygen Saturation (mmHg) Body Weight (kg) Temperature (C) | Supine<br>Supine<br>Supine<br>Supine | XXX +<br>XXX<br>XXX<br>XXX<br>XXX<br>XXX<br>XXX.X | |
| | C1 TRT D2 | DDMMMYYYY HH:MM | XXX | Pulse Rate (bpm) Respiratory Rate (bpm) Systolic BP (mmHg) Diastolic BP (mmHg) Oxygen Saturation (mmHg) Body Weight (kg) Temperature (C) | Supine<br>Supine<br>Supine<br>Supine | XXX +<br>XXX<br>XXX<br>XXX<br>XXX<br>XXX.X<br>XX.X | XX<br>XX<br>XX<br>XX<br>XX<br>XX<br>X.X |

<repeat for Day 3, Day 4, Day 5, Day 6 and Day 10 visits of Cycle 1>
<for Cycle 2 to last-1 cycle, repeat from Day 1 to Day 6 visits if relevant>
<for the last cycle, repeat also for Day 22 visit and Day 28 follow-up visit>

Study Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY. Baseline was the last non-missing assessment prior or on the first dose.

+ Results of clinical importance (see SAP). BP = Blood Pressure; bpm = beats per minute; ND = Not Done.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM) Filename: (Specify file name.rtf)

#### PROGRAMMING NOTES:

• Repeat for all doses groups



Sponsor: CicloMed Protocol: CPX-POM-001

Statistical Analysis Plan

(TFL shells):


Protocol: CPX-POM-001 --- DELIVERY TYPE ---- Page 1 of X

Listing 16.2.8-6 - ECG Results and Interpretation (All Patients)

CPX-POM Dose Group: 30 mg/m^2

| Center/<br>Patient | Visit | Assessment Date (Day) | Parameter (unit) | Clinician Interpretation | Result | Change<br>from<br>baseline |
|---|---|---|---|---|---|---|
| XXXX | BAS | DDMMMYYYY (XXX) | Heart Rate (bpm) PR interval (msec) QRS duration (msec) QT interval (msec) QTcB interval (msec) QTcF interval (msec) | Normal<br>Normal<br>Normal<br>Normal<br>Normal | XXX | |
| | C1 TRT D5 | DDMMMYYYY (XXX) | Heart Rate (bpm) PR interval (msec) QRS duration (msec) QT interval (msec) QTcB interval (msec) QTcF interval (msec) | Abnormal, Clinical Significant Normal Normal Normal Abnormal, Not Clinical Significant Abnormal, Not Clinical Significant | XXX ++<br>XXX +<br>XXX + | XX * |

<for Cycle 2 to last-1 cycle, repeat for Day 1 visit if relevant> <for the last cycle, repeat also for Day 28 follow-up visit>

Day was from the date of first dose of CPX-POM administration. Dates are displayed as DDMMMYYYY. Baseline was the last non-missing assessment prior or on the first dose date.

Filename: (Specify file name.rtf)

QTcB and QTcF: +: >450 msec; ++: > 480 msec; +++: >500 msec; \*: > 30 msec above baseline; \*\*: > 60 msec above baseline. R = repeated/ unscheduled assessment.

Program: (Program name.sas) (run on: DDMMMYYYY HH:MM)

#### PROGRAMMING NOTES:

• Repeat for all dose groups.